CLINICAL TRIAL: NCT07167628
Title: Neurological Complications and Intensive-Care Workload After Emergency Repair of Acute Type A Aortic Dissection: A Retrospective Cohort Study
Brief Title: Neurological Complications and ICU Workload After Emergency Repair of Acute Type A Aortic Dissection
Acronym: ATAAD-ICU
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH114-REC1-139
Record Dates: First submitted 2025-08-31; First posted 2025-09-11 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Aortic Dissection; Stroke; Paraplegia; AKI - Acute Kidney Injury; Coma; Delirium
Keywords: Acute type A aortic dissection; Neurological complications; Intensive care unit; ICU workload; ICU length of stay; Mechanical ventilation; Hospital length of stay; Retrospective cohort; Nursing workload; Taiwan
MeSH Terms: conditions — Aortic Dissection; Stroke; Paraplegia; Acute Kidney Injury; Coma; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults undergoing emergency ATAAD repair: Single-center retrospective cohort of consecutive adults (≥18 years) who underwent emergency repair of acute type A aortic dissection at China Medical University Hospital between 2021-01-01 and 2025-04-30; all participants are pooled into one cohort with no protocol-assigned interventions; outcomes are obtained from de-identified records to assess neurological complications and ICU resource use.

SUMMARY:
Single-center retrospective cohort at China Medical University Hospital (Taichung, Taiwan) using fully de-identified electronic health records. Consecutive adults who underwent emergency repair of acute type A aortic dissection between 2021-01-01 and 2025-04-30 were pooled into one cohort. The study measures the incidence and patterns of early postoperative neurological complications and evaluates their association with intensive care unit (ICU) resource use, focusing on prolonged ICU length of stay (LOS ≥ 10 days), ICU and hospital LOS, and duration of mechanical ventilation (MV). No new data collection or patient contact occurs. Institutional Review Board (IRB) approval: CMUH114-REC1-139.

DETAILED DESCRIPTION:
Adults (≥ 18 years) undergoing emergency repair for acute type A aortic dissection (ATAAD) at China Medical University Hospital (CMUH) during 2021-01-01 to 2025-04-30 were screened. Exclusions: missing key variables, preoperative stroke within 30 days or modified Rankin Scale (mRS) ≥ 4, pregnancy. The analytic cohort included 274 of 309 screened patients. Neurological complications comprise radiology-confirmed stroke, other focal neurological deficits, paraplegia, or sustained coma/encephalopathy recorded by neurology consultation. Prolonged ICU stay is prespecified as ICU LOS ≥ 10 days in the index admission. Outcomes: primary outcomes are prolonged ICU stay and any postoperative neurological complication; secondary outcomes are ICU LOS (days), duration of mechanical ventilation (hours), hospital LOS (days), in-hospital mortality, and in-hospital death within 30 days of the index surgery. Analyses are performed in R version 4.5.1. Continuous variables are summarized as medians with interquartile ranges (IQRs) and compared using the Mann-Whitney U test; categorical variables are presented as counts and percentages and compared using chi-square or Fisher exact tests. Multivariable logistic regression identifies factors associated with prolonged ICU stay (ICU LOS ≥ 10 days) among hospital survivors using a priori covariates (age, sex, chronic kidney disease stage 4-5, operation time, cardiopulmonary bypass [CPB] time, intraoperative red blood cell [RBC] units transfused, postoperative acute kidney injury [AKI], any postoperative neurological complication). A prespecified sensitivity analysis in the full cohort treats the endpoint as ICU LOS ≥ 10 days or in-hospital death using the same prespecified covariates. Data were de-identified before analysis and stored on secure hospital servers; the study is minimal risk and does not involve United States Food and Drug Administration (US FDA) regulated products.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) who underwent emergency repair of acute type A aortic dissection at China Medical University Hospital between 2021-01-01 and 2025-04-30.

Exclusion Criteria:

* Missing data in key variables required for analyses.
* Preoperative ischemic stroke within 30 days before surgery or preoperative modified Rankin Scale ≥4.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adults undergoing emergency repair of acute type A aortic dissection at a single tertiary centre ICU in Taichung, Taiwan (2021-01-01 to 2025-04-30).
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Prolonged ICU length of stay (LOS ≥10 days) | Through ICU discharge during the index admission (up to 30 days).
  Proportion of participants with ICU LOS ≥10 days during the index ICU admission. Unit of measure: percent.
Any postoperative neurological complication | Through hospital discharge during the index admission (up to 30 days).
  Proportion with stroke (CT/MRI confirmed), other focal neurological deficits, paraplegia, or sustained coma/encephalopathy recorded by neurology consultation. Unit of measure: percent.

SECONDARY OUTCOMES:
ICU length of stay (days) | Through ICU discharge during the index admission (up to 30 days).
  ICU LOS summarized as median and IQR; larger values indicate greater resource use. Unit of measure: days.
Duration of mechanical ventilation (hours) | Through final extubation during the index hospitalization (up to 40 days).
  Cumulative hours of invasive ventilation from ICU arrival to final extubation. Unit of measure: hours.
Hospital length of stay (days) | Through hospital discharge during the index admission (up to 65 days).
  Days from hospital admission to discharge; deaths counted up to date of death. Unit of measure: days.
In-hospital mortality | Through hospital discharge during the index admission (up to 30 days).
  All-cause death before discharge from the index hospitalization. Unit of measure: percent.
In-hospital mortality within 30 days | Up to 30 days after index surgery, during the index hospitalization.
  All-cause death occurring during the index hospitalization within 30 days after the index surgery (deaths after hospital discharge were not captured).

CONTACTS AND LOCATIONS:
Overall Officials: En-Bo Wu, MD, Principal Investigator — Department of Anesthesiology, China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taichung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. The dataset consists of de-identified electronic health records governed by CMUH institutional policy and IRB approval (CMUH114-REC1-139), which restrict external transfer. Aggregate results or summary tables may be provided on reasonable request, subject to additional REC approval and data-use agreements.

REFERENCES:
- [Background] Vandenbroucke JP, von Elm E, Altman DG, Gotzsche PC, Mulrow CD, Pocock SJ, Poole C, Schlesselman JJ, Egger M; STROBE Initiative. Strengthening the Reporting of Observational Studies in Epidemiology (STROBE): explanation and elaboration. PLoS Med. 2007 Oct 16;4(10):e297. doi: 10.1371/journal.pmed.0040297. PMID 17941715
- [Background] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Background] Sacco RL, Kasner SE, Broderick JP, Caplan LR, Connors JJ, Culebras A, Elkind MS, George MG, Hamdan AD, Higashida RT, Hoh BL, Janis LS, Kase CS, Kleindorfer DO, Lee JM, Moseley ME, Peterson ED, Turan TN, Valderrama AL, Vinters HV; American Heart Association Stroke Council, Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular and Stroke Nursing; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Council on Nutrition, Physical Activity and Metabolism. An updated definition of stroke for the 21st century: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Jul;44(7):2064-89. doi: 10.1161/STR.0b013e318296aeca. Epub 2013 May 7. PMID 23652265
- [Background] Queijo AF, Martins RS, Andolhe R, Oliveira EM, Barbosa RL, Padilha KG. Nursing workload in neurological intensive care units: cross-sectional study. Intensive Crit Care Nurs. 2013 Apr;29(2):112-6. doi: 10.1016/j.iccn.2012.08.001. Epub 2012 Sep 19. PMID 22999497
- [Background] Branch-Elliman W, Wright SB, Gillis JM, Howell MD. Estimated nursing workload for the implementation of ventilator bundles. BMJ Qual Saf. 2013 Apr;22(4):357-61. doi: 10.1136/bmjqs-2012-001372. Epub 2013 Feb 21. PMID 23431219
- [Background] Lewis K, Balas MC, Stollings JL, McNett M, Girard TD, Chanques G, Kho ME, Pandharipande PP, Weinhouse GL, Brummel NE, Chlan LL, Cordoza M, Duby JJ, Gelinas C, Hall-Melnychuk EL, Krupp A, Louzon PR, Tate JA, Young B, Jennings R, Hines A, Ross C, Carayannopoulos KL, Aldrich JM. A Focused Update to the Clinical Practice Guidelines for the Prevention and Management of Pain, Anxiety, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2025 Mar 1;53(3):e711-e727. doi: 10.1097/CCM.0000000000006574. Epub 2025 Feb 21. PMID 39982143
- [Background] Liu H, Zhang S, Zhang C, Gao Q, Liu Y, Liao F, Ge S. Risk factors for prolonged postoperative ICU stay in the patients with Stanford type A aortic dissection. J Cardiothorac Surg. 2024 Feb 3;19(1):46. doi: 10.1186/s13019-024-02548-7. PMID 38310273
- [Background] Dumfarth J, Kofler M, Stastny L, Plaikner M, Krapf C, Semsroth S, Grimm M. Stroke after emergent surgery for acute type A aortic dissection: predictors, outcome and neurological recovery. Eur J Cardiothorac Surg. 2018 May 1;53(5):1013-1020. doi: 10.1093/ejcts/ezx465. PMID 29360972
- [Background] Biancari F, Herve A, Peterss S, Radner C, Buech J, Pettinari M, Rodriguez Lega J, Pinto AG, Fiore A, Onorati F, Francica A, Wisniewski K, Demal T, Conradi L, Rocek J, Kacer P, Gatti G, Vendramin I, Rinaldi M, Ferrante L, Pruna-Guillen R, Quintana E, DI Perna D, Mariscalco G, Jormalainen M, Field M, Harky A, Dell'aquila AM, Juvonen T, Makikallio T, Perrotti A. Predictors, prognosis and costs of prolonged intensive care unit stay after surgery for type A aortic dissection. Minerva Anestesiol. 2024 Jul-Aug;90(7-8):654-661. doi: 10.23736/S0375-9393.24.18210-7. PMID 39021141
- [Background] Arabi YM, Phua J, Koh Y, Du B, Faruq MO, Nishimura M, Fang WF, Gomersall C, Al Rahma HN, Tamim H, Al-Dorzi HM, Al-Hameed FM, Adhikari NK, Sadat M; Asian Critical Care Clinical Trials Group. Structure, Organization, and Delivery of Critical Care in Asian ICUs. Crit Care Med. 2016 Oct;44(10):e940-8. doi: 10.1097/CCM.0000000000001854. PMID 27347762